CLINICAL TRIAL: NCT05422729
Title: A Multidisciplinary-led Personalised mHealth-supported Coach for Reducing Midlife Stroke Risk
Brief Title: mHealth-supported Coach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Helen YL Chan, Associate Professor (Dr), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 05200218
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Heart Disease Risk Factors
Keywords: Primary Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalised mHeatlh-supported coaching programme (Experimental): Three monthly individual consultation session, supported with a specific mobile application.
  Interventions: Behavioral: mHealth-supported coaching
- Traditional in-person health coaching programme (Active Comparator): Three monthly individual consultation sessions.
  Interventions: Behavioral: Conventional Health coaching

INTERVENTIONS:
Behavioral: mHealth-supported coaching — The intervention includes two components. Three individual consultation sessions based on a health coaching protocol developed by a multidisciplinary team. A mobile application provides educational information about healthy lifestyles, knowledge quizzes, telemonitoring function and virtual platform for sharing.
  Arms: Personalised mHeatlh-supported coaching programme
Behavioral: Conventional Health coaching — Three individual consultation sessions delivered by a nurse.
  Arms: Traditional in-person health coaching programme

SUMMARY:
A randomised controlled trial to evaluate the effects of a personalised mHealth-supported coach programme in the middle-aged group with stroke risk.

DETAILED DESCRIPTION:
Aim: To evaluate the effects of a personalised mHealth-supported coach programme on the adoption of health-promoting behaviours in the middle-aged group, in comparison with usual care.

Design: A 24-month prospective two-arm, parallel-group, single-blinded, repeated-measure randomised controlled trial will be conducted.

Participants: People who aged between 40 and 64, mentally competent, have a non-laboratory INTERHEART risk score (IHRS) of 10 or higher, communicable in Chinese and free from stroke and transient ischemic attack (TIA) or other cardiovascular disease will be eligible to the study. A total of 164 participants will be recruited through a district community centre and randomly assigned on 1:1 ratio to the intervention group or the control group.

Intervention: A theory-based mHealth-supported coach programme, including individual consultation sessions and a mobile application with a virtual sharing platform, is developed by a multidisciplinary team for the intervention group over three months, whereas the control group receives usual care.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnic
* able to read Chinese and communicate in Cantonese/Mandarin
* with non-laboratory IHRS score 10 or higher

Exclusion Criteria:

* mentally incompetent
* previously diagnosed with stroke, TIA, MI, coronary heart disease, heart failure or atrial fibrillation
* with eye or retinal disease
* with terminal disease with an expected life expectancy less than six months
* being pregnant
* have enrolled in other lifestyle-based or exercise-based projects
* do have mobile devices or internet service to access the mobile application

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-04 (Estimated)

PRIMARY OUTCOMES:
Health-promoting behaviours | 3-month post-allocation
  Four subscales, including health responsibility, nutrition, physical activity and stress management, of the Health Promoting Lifestyle Profile II. The possible score range from 34 to 136, with a higher score meaning healthier lifestyles were adopted.
Health-promoting behaviours | 6-month post-allocation
  Four subscales, including health responsibility, nutrition, physical activity and stress management, of the Health Promoting Lifestyle Profile II. The possible score range from 34 to 136, with a higher score meaning healthier lifestyles were adopted.

SECONDARY OUTCOMES:
Self-efficacy of adopting health-promoting behaviours | 3-month post-allocation
  The adapted version of the Diabetes Mellitus Type II Self Efficacy Scale will be used. Participants will rate their level of confidence in various behaviours, in diet control, weight control and lifestyle management, by using a five-point Likert scale. The possible scores ranged from 7 to 35, with a higher score meaning a higher level of self-efficacy.
Self-efficacy | 6-month post-allocation
  The adapted version of the Diabetes Mellitus Type II Self Efficacy Scale will be used. Participants will rate their level of confidence in various behaviours, in diet control, weight control and lifestyle management, by using a five-point Likert scale. The possible scores ranged from 7 to 35, with a higher score meaning a higher level of self-efficacy.
INTERHEART risk score | 3-month post-allocation
  The score was calculated based on the weighted sum of nine risk factors, including age, sex, lifestyles and psychosocial wellbeing, which were significantly related to cardiovasuclar diseases. The possible score range was 0 - 48, in which a higher score corresponds to higher risk.
INTERHEART risk score | 6-month post-allocation
  The score was calculated based on the weighted sum of nine risk factors, including age, sex, lifestyles and psychosocial wellbeing, which were significantly related to cardiovasuclar diseases. The possible score range was 0 - 48, in which a higher score corresponds to higher risk.
automatic retinal image analysis | 3-month post-allocation
  Retinal fundus image will be obtained from both eyes of the participant using a non-mydriatic digital retinal camera (Canon CR-2 AF, U.S.A., Inc). Stroke risk estimation will be determined through fractural analysis, statistical texture analysis and high-order spectra analysis based on the retinal vessel parameters. The ARIA-stroke algorithm developed using R and Matlab software has a sensitivity and a specificity of 94.7% and 100%, respectively. The value between 0.5 and 0.7 is considered as moderate risk, while high risk is considered at 0.7 or higher.
automatic retinal image analysis (ARIA) | 6-month post-allocation
  Retinal fundus image will be obtained from both eyes of the participant using a non-mydriatic digital retinal camera (Canon CR-2 AF, U.S.A., Inc). Stroke risk estimation will be determined through fractural analysis, statistical texture analysis and high-order spectra analysis based on the retinal vessel parameters. The ARIA-stroke algorithm developed using R and Matlab software has a sensitivity and a specificity of 94.7% and 100%, respectively. The value between 0.5 and 0.7 is considered as moderate risk, while high risk is considered at 0.7 or higher.
Psychological distress | 3-month post-allocation
  The Depression Anxiety Stress Scale (DASS-21)includes 21 items, with 7 in each subscale: depression, anxiety and stress. Participants will rate their level of agreement with the statements on a 4-point Likert scale, from 0 (not apply to me at all) to 3 (applied to me very much). The potential scores range from 0 to 63, with a higher score means higher level of distress experienced.
Psychological distress | 6-month post-allocation
  The Depression Anxiety Stress Scale (DASS-21)includes 21 items, with 7 in each subscale: depression, anxiety and stress. Participants will rate their level of agreement with the statements on a 4-point Likert scale, from 0 (not apply to me at all) to 3 (applied to me very much). The potential scores range from 0 to 63, with a higher score means higher level of distress experienced.
Change in Blood pressure | Between baseline and 3-month post-allocation
  Blood pressure measurement will be carried out, after 10 min of rest, on the left arm in a sitting posture by using an electronic sphygmomanometer.
Change in Blood pressure | Between 3-month and 6-month post-allocation
  Blood pressure measurement will be carried out, after 10 min of rest, on the left arm in a sitting posture by using an electronic sphygmomanometer.
Change in Body mass index (BMI) | Between baseline and 3-month post-allocation
  BMI will be calculated by dividing the weight (in kilogram) by the height (in meter) squared. The height will be measured using a stadiometer, and body weight will be measured using an electronic scale.
Change in Body mass index(BMI) | Between 3-month and 6-month post-allocation
  BMI will be calculated by dividing the weight (in kilogram) by the height (in meter) squared. The height will be measured using a stadiometer, and body weight will be measured using an electronic scale.
Change in Waist-hip ratio (WHR) | Between baseline and 3-month post-allocation
  WHR will be used for determining body fat distribution. Waist circumference will be measured at the mid-point between the lowest rib and the iliac crest, whereas hip circumference will be measured at the widest level over the great trochanters. The two measurements will be measured to the nearest 0.1 cm by using a measuring tape.
Change in Waist-hip ratio (WHR) | Between 3-month and 6-month post-allocation
  WHR will be used for determining body fat distribution. Waist circumference will be measured at the mid-point between the lowest rib and the iliac crest, whereas hip circumference will be measured at the widest level over the great trochanters. The two measurements will be measured to the nearest 0.1 cm by using a measuring tape.
Change in Fasting blood glucose | Between baseline and 3-month post-allocation
  Blood samples will be taken by an experienced nurse and sent to accredited commercial biochemistry laboratories for analysis.
Change in Fasting blood glucose | Between 3-month and 6-month post-allocation
  Blood samples will be taken by an experienced nurse and sent to accredited commercial biochemistry laboratories for analysis.
Change in Blood lipid profile | Between baseline and 3-month post-allocation
  The profile includes ncluding triglyceride, total Cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C). Blood samples will be taken by an experienced nurse and sent to accredited commercial biochemistry laboratories for analysis.
Change in Blood lipid profile | Between 3-month and 6-month post-allocation
  The profile includes ncluding triglyceride, total Cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C). Blood samples will be taken by an experienced nurse and sent to accredited commercial biochemistry laboratories for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Y Chan, Ph.D, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided